CLINICAL TRIAL: NCT06320613
Title: Effect of Using Snap-Needle Therapy in Combination With Ginger Paste During Anesthesia Recovery on the Recovery of Gastrointestinal Function After Gynecologic Laparoscopy
Brief Title: Effect of Implementing Snap-needle Therapy Combined With Ginger Paste During Anesthesia Recovery on the Recovery of Gastrointestinal Function After Gynecologic Laparoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weifang Medical University (Other)
Collaborators: Weifang People's Hospital (Other)
Responsible Party: Principal Investigator, Lin Cheng, Pricipal Investigator, Weifang Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KYLL20240117-2
Record Dates: First submitted 2024-03-01; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Motility; Postoperative Nausea and Vomiting
Keywords: Gastrointestinal Motility; Recovery of Function; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group acupuncture(snap-needle) (Active Comparator): Patients in the acupuncture group received acupuncture therapy (snap-needle therapy) for 24 hours. Results of the study were collected at six assessment periods of 0-0.5 h, 0-1 h, 1-3 h, 4-6h, 6-12 h, and 12-24 h after anesthesia. Conducted by an independent researcher.
  Interventions: Other: Acupuncture therapy
- Experimental Ginger (Active Comparator): Patients in the Ginger Acupuncture Point Patch group received ginger patch therapy and the ginger patch was removed within 6h. Study results were collected at six assessment periods of 0-0.5h, 0-1h, 1-3h, 4-6h, 6-12h, and 12-24h after anesthesia. Conducted by an independent researcher.
  Interventions: Other: Ginger Acupuncture Point Patch
- Experimental group Acupuncture combined with ginger (Active Comparator): Patients in the Acupuncture combined with ginger group received acupuncture treatment (snap-needle therapy) combined with ginger compresses, which were removed within 6h and snap-needles were removed after 24 hours. Study results were collected at six assessment periods of 0-0.5h, 0-1h, 1-3h, 4-6h, 6-12h, and 12-24h after anesthesia. Conducted by an independent researcher.
  Interventions: Other: Acupuncture therapy; Other: Ginger Acupuncture Point Patch

INTERVENTIONS:
Other: Acupuncture therapy — After disinfecting (alcohol or 0.9% Normal saline) the skin at the acupuncture point, use small tweezers to clip the handle of the needle, remove the adhesive tape and stab the acupuncture point at a perpendicular angle, and then press the thumb with moderate pressure on the snap-needle embedded needle site in order for the patient to feel localized soreness and distension as appropriate. The snap-needle was removed after 24 hours, and the pressing time point remained unchanged.
  Other Names: Qin acupuncture therapy; snap-needle therapy
  Arms: Experimental group Acupuncture combined with ginger; Experimental group acupuncture(snap-needle)
Other: Ginger Acupuncture Point Patch — Ginger was thinly sliced and then cut into 2-3cm diameter ginger discs according to a circular mold and covered with a sterile circular dressing. The ginger compress was removed within 6 hours.
  Arms: Experimental Ginger; Experimental group Acupuncture combined with ginger

SUMMARY:
The aim of this study was to investigate the effect of implementing snap-needle therapy combined with ginger paste during anesthesia recovery on the recovery of gastrointestinal function after gynecological laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I or II;
2. Performing gynecologic laparoscopic procedures under general anesthesia;

Exclusion Criteria:

1. Age ≤ 18 or ≥65;
2. The patient has a previous history of PONV, digestive disorders, etc;
3. Ulcers, infections, and skin tears at acupressure and acupuncture (snap-needle) treatment sites;
4. Patients allergic to ginger；
5. Inability to follow protocol or refusal to participant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | Measured at 0.5 hours postoperatively.
  The Index of Nausea and Vomiting and Retching (INVR) was used in this study. The scale consists of 8 items with 3 dimensions, which can quantify the number of occurrences, duration and severity of symptoms. The scale is scored using the Likert method, with a total of 32 points on a 5-point scale ranging from 0 to 4. The higher the score, the more severe the symptoms of nausea, vomiting, and dry heaving (entries 1, 6, and 7 are reverse scored). According to the score, nausea, vomiting and dry heaving symptoms can be categorized into five grades: 0, I, II, III and IV, and grade ≥I means that the symptom occurs. The severity and incidence of PONV at 0.5 hours postoperatively.
Postoperative nausea and vomiting | Measured at 1 hours postoperatively.
  The Index of Nausea and Vomiting and Retching (INVR) was used in this study. The scale consists of 8 items with 3 dimensions, which can quantify the number of occurrences, duration and severity of symptoms. The scale is scored using the Likert method, with a total of 32 points on a 5-point scale ranging from 0 to 4. The higher the score, the more severe the symptoms of nausea, vomiting, and dry heaving (entries 1, 6, and 7 are reverse scored). According to the score, nausea, vomiting and dry heaving symptoms can be categorized into five grades: 0, I, II, III and IV, and grade ≥I means that the symptom occurs. The severity and incidence of PONV at 1 hours postoperatively.
Postoperative nausea and vomiting | Measured at 3 hours postoperatively.
  The Index of Nausea and Vomiting and Retching (INVR) was used in this study. The scale consists of 8 items with 3 dimensions, which can quantify the number of occurrences, duration and severity of symptoms. The scale is scored using the Likert method, with a total of 32 points on a 5-point scale ranging from 0 to 4. The higher the score, the more severe the symptoms of nausea, vomiting, and dry heaving (entries 1, 6, and 7 are reverse scored). According to the score, nausea, vomiting and dry heaving symptoms can be categorized into five grades: 0, I, II, III and IV, and grade ≥I means that the symptom occurs. The severity and incidence of PONV at 3 hours postoperatively.
Postoperative nausea and vomiting | Measured at 6 hours postoperatively.
  The Index of Nausea and Vomiting and Retching (INVR) was used in this study. The scale consists of 8 items with 3 dimensions, which can quantify the number of occurrences, duration and severity of symptoms. The scale is scored using the Likert method, with a total of 32 points on a 5-point scale ranging from 0 to 4. The higher the score, the more severe the symptoms of nausea, vomiting, and dry heaving (entries 1, 6, and 7 are reverse scored). According to the score, nausea, vomiting and dry heaving symptoms can be categorized into five grades: 0, I, II, III and IV, and grade ≥I means that the symptom occurs. The severity and incidence of PONV at 6 hours postoperatively.
Postoperative nausea and vomiting | Measured at 12 hours postoperatively.
  The Index of Nausea and Vomiting and Retching (INVR) was used in this study. The scale consists of 8 items with 3 dimensions, which can quantify the number of occurrences, duration and severity of symptoms. The scale is scored using the Likert method, with a total of 32 points on a 5-point scale ranging from 0 to 4. The higher the score, the more severe the symptoms of nausea, vomiting, and dry heaving (entries 1, 6, and 7 are reverse scored). According to the score, nausea, vomiting and dry heaving symptoms can be categorized into five grades: 0, I, II, III and IV, and grade ≥I means that the symptom occurs. The severity and incidence of PONV at 12 hours postoperatively.
Postoperative nausea and vomiting | Measured at 24 hours postoperatively.
  The Index of Nausea and Vomiting and Retching (INVR) was used in this study. The scale consists of 8 items with 3 dimensions, which can quantify the number of occurrences, duration and severity of symptoms. The scale is scored using the Likert method, with a total of 32 points on a 5-point scale ranging from 0 to 4. The higher the score, the more severe the symptoms of nausea, vomiting, and dry heaving (entries 1, 6, and 7 are reverse scored). According to the score, nausea, vomiting and dry heaving symptoms can be categorized into five grades: 0, I, II, III and IV, and grade ≥I means that the symptom occurs. The severity and incidence of PONV at 24 hours postoperatively.
Abdominal distention | Measured at 0.5 hours postoperatively.
  The severity and incidence of Abdominal distention at 0.5 hours postoperatively.
Abdominal distention | Measured at 1 hours postoperatively.
  The severity and incidence of Abdominal distention at 1 hours postoperatively.
Abdominal distention | Measured at 3 hours postoperatively.
  The severity and incidence of Abdominal distention at 3 hours postoperatively.
Abdominal distention | Measured at 6 hours postoperatively.
  The severity and incidence of Abdominal distention at 6 hours postoperatively.
Abdominal distention | Measured at 12 hours postoperatively.
  The severity and incidence of Abdominal distention at 12 hours postoperatively.
Abdominal distention | Measured at 24 hours postoperatively.
  The severity and incidence of Abdominal distention at 24 hours postoperatively.
Time to first flatus | Approximately 24 hours after surgery.
  Record the time of the first flatus. The earlier the time of first flatus, the earlier the time of recovery of gastrointestinal function.

SECONDARY OUTCOMES:
Postoperative pain response | Measured at 0.5 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 0.5 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Postoperative pain response | Measured at 1 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 1 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Postoperative pain response | Measured at 3 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 3 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Postoperative pain response | Measured at 6 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 6 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Postoperative pain response | Measured at 12 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 12 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Postoperative pain response | Measured at 24 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 24 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Consumption of postoperative analgesic | Approximately 24 hours after surgery.
  Record the type and dosage of postoperative analgesic within 24 hours after surgery.
Consumption of postoperative rescue antiemetic | Approximately 24 hours after surgery
  Record the type and dosage of postoperative rescue antiemetic within 24 hours after surgery.
Time to first defecation | Approximately 24 hours after surgery.
  Record the time of first defecation.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Cheng, B.S, Principal Investigator — Weifang People's Hospital
Locations (1):
- Lin Cheng, Weifang, Shandong, China

IPD SHARING:
Plan to Share IPD: No